CLINICAL TRIAL: NCT05968131
Title: Comparative Effects of Proprioceptive Training and Routine Physical Therapy on Balance and Quality Of Life in Individuals With Diabetic Peripheral Neuropathy
Brief Title: Comparative Effects of Proprioceptive Training and Routine Physical Therapy on Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Sidra Naz, Principal Investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/997/2021
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetes; Diabetic Peripheral Neuropathy; Balance; Quality of Life; Proprioceptive Training; Physiotherapy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study will be single-blinded. The assessor will be unaware of the treatment given to both groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physical Therapy (Active Comparator): Conventional Physical Therapy will consist of application heat pack, ROM exercises, stretching, and strengthening exercises
  Interventions: Other: Conventional Physical Therapy
- Conventional Physical Therapy with Proprioceptive Training Exercises (Experimental): Conventional Physical Therapy with Proprioceptive Training Exercises
  Interventions: Other: Conventional Physical Therapy; Other: Conventional Physical Therapy with Proprioceptive Training Exercises

INTERVENTIONS:
Other: Conventional Physical Therapy — The control group will receive only strength training intervention included the following components:
  Range Of Motion Exercises: movements to the extent possible of the knee (flexion-extension), ankle (dorsi-plantar flexion), forefoot (inversion-eversion) and toe (flexion-extension).
  5 repetitions of each ROM exercise will be done for 2 minutes. Muscle Strengthening Exercises: active movements against resistance (using a Thera band) at the knee (flexion-extension), ankle (dorsi-plantar flexion), forefoot (inversion- eversion) and toe (flexion-extension).
  Each Strengthening exercise will be performed for 5 minutes with 10 repetitions.
Other: Conventional Physical Therapy with Proprioceptive Training Exercises — Interventional group will receive strengthening intervention as well as proprioceptive training for 32 sessions. ROM and Strengthening exercise will be performed same as in control group.
  Exercises For Proprioceptive Training: Intervention group will practice an additional 24 minutes of proprioceptive training (two minutes rest prior to performing this training). A circuit with different floor texture composed of 6 stations of exercises to stimulate the sole of foot where participant had to improve gait by stepping with alternate feet marker placed on ground and progression will be done by modify the speed and direction. Material used to build the circuit are in following order: 10 cm thick foam, a wood box with beans, a 2 cm thick mat with density lower than foam, a wooden box filled with sand, balance board to train the lateral balance reactions, a wooden box filled with cotton. Duration of this training is 24 minutes; patient will spend 4 minutes on each station.
  Arms: Conventional Physical Therapy with Proprioceptive Training Exercises

SUMMARY:
This project will compare the effects of proprioceptive training with routine physical therapy intervention on improving balance and health-related quality of life in individuals with diabetic neuropathy. The subjects who met the inclusion/exclusion criteria will be allocated for controlled and experimental groups. Subjects will be selected from the outpatient clinic of the Department of Physical Therapy. Subjects will be divided randomly into two equal groups. The study will be single-blinded. Subjects will be randomized into two groups Group A & Group B.Baseline data will be collected then collect data at2nd, 4th Week and 8th week.Individuals will be assigned to the intervention group receive proprioceptive training and strengthening interventions guided by a physiotherapist for 8 weeks. Session will begin with a 5 min pre-exercise warm-up of gentle stretches and will be ended with a 5 min cool-down of slow walking. Participant should encourage to perform the exercises for at least four times a week and home-based exercises for once a day.

DETAILED DESCRIPTION:
This project will compare the effects of proprioceptive training with routine physical therapy intervention on improving balance and health-related quality of life in individuals with diabetic neuropathy. The subjects who met the inclusion/exclusion criteria will be allocated for controlled and experimental groups. Subjects will be selected from the outpatient clinic of the Department of Physical Therapy. Subjects will be divided randomly into two equal groups. The study will be single-blinded. Subjects will be randomized into two groups Group A & Group B.Baseline data will be collected then collect data at2nd, 4th Week, and 8th weeks.

FOR CONVENTIONAL PHYSICAL THERAPY GROUPS:

The control group will receive only strength training intervention included the following components:

Range Of Motion Exercises: movements to the extent possible of the knee (flexion-extension), ankle (Dorsi, plantar flexion), forefoot (inversion-eversion), and toe (flexion-extension).

5 repetitions of each ROM exercise will be done for 2 minutes. Muscle Strengthening Exercises: active movements against resistance (using a Thera band) at the knee (flexion-extension), ankle (dorsiflexion and plantar flexion), forefoot (inversion- eversion), and toe (flexion-extension).

Each Strengthening exercise will be performed for 5 minutes with 10 repetitions.

FOR INTERVENTIONAL PHYSICAL THERAPY GROUP:

The interventional group will receive strengthening intervention as well as proprioceptive training for 32 sessions. ROM and Strengthening exercises will be performed the same as in the control group.

Exercises For Proprioceptive Training: Intervention group will practice an additional 24 minutes of proprioceptive training (two minutes rest prior to performing this training). A circuit with different floor textures composed of 6 stations of exercises to stimulate the sole of the foot where the participant had to improve gait by stepping with alternate feet marker placed on the ground and progression will be done by modifying the speed and direction. The material used to build the circuit are in the following order: 10 cm thick foam, a wood box with beans, a 2 cm thick mat with density lower than foam, a wooden box filled with sand, a balance board to train the lateral balance reactions, a wooden box filled with cotton. The duration of this training is 24 minutes; the patient will spend 4 minutes on each station

ELIGIBILITY:
Inclusion Criteria:

1. Age is between 35- 65 years
2. Both gender (male & female)
3. Diagnosed Type 2 Diabetes with the appearance of peripheral neuropathy from at least six month
4. Michigan Neuropathy Screening Instrument Questionnaire score of 5 or greater.
5. Patient is able to stand on both feet

Exclusion Criteria:

1. Foot ulceration/ Infection
2. Amputation
3. Inner ear infection
4. Neurological illness that affects balance
5. Musculoskeletal problems such as vertebral column and limb deformity
6. Patient with any orthotic device

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Balance Score | The balance score will be monitored at baseline at the recruitment in the study, at 4th week and 8th week of intervention.
  Berg Balance Scale (BBS) evaluates functional balance before and after intervention. It is a valid and reliable scale including 14 functional tests, which can quantitatively evaluate balance in community dwelling adults and patients with balance disorders. Berg Balance Scale completion needs 10-20 min. and its score represents the participant's ability to control postural balance. It score ranges from 0 to 56. A total score of 0-20 reflects mobility by wheelchair, 21 to 40 walking with assistance, and a score of 41 to 56 walking independently.
Change in Quality of Life | Quality of life will be measured at the baseline, and any change in quality of life will be measured at 4th week and 8th week of intervention.
  It is defined by the World Health Organization as individual's perception of their position in life in the context of the culture and value systems in which they live, and in relation to their goals, expectations, standards and concerns.33The 36-Item Short Form Health Survey questionnaire (SF-36) is popular instrument for evaluating Health-Related Quality of Life. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Component analyses showed that there are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS). All scales do contribute in different proportions to the scoring of both PCS and MCS measures. It scores range from 0 to 100, with higher scores representing better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Naz, MS, Principal Investigator — University of Lahore
Locations (1):
- District Head Quarter Hospital Layyah., Layyah, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sendi RA, Mahrus AM, Saeed RM, Mohammed MA, Al-Dubai SAR. Diabetic peripheral neuropathy among Saudi diabetic patients: A multicenter cross-sectional study at primary health care setting. J Family Med Prim Care. 2020 Jan 28;9(1):197-201. doi: 10.4103/jfmpc.jfmpc_927_19. eCollection 2020 Jan. PMID 32110590
- [Background] Riandini T, Khoo EYH, Tai BC, Tavintharan S, Phua MSLA, Chandran K, Hwang SW, Venkataraman K. Fall Risk and Balance Confidence in Patients With Diabetic Peripheral Neuropathy: An Observational Study. Front Endocrinol (Lausanne). 2020 Oct 23;11:573804. doi: 10.3389/fendo.2020.573804. eCollection 2020. PMID 33193090
- [Background] Feldman EL, Nave KA, Jensen TS, Bennett DLH. New Horizons in Diabetic Neuropathy: Mechanisms, Bioenergetics, and Pain. Neuron. 2017 Mar 22;93(6):1296-1313. doi: 10.1016/j.neuron.2017.02.005. PMID 28334605